CLINICAL TRIAL: NCT07333651
Title: Standard-of-Care Systemic Therapy With or Without Image-Guided 125I Seed Implantation in Patients With Oligoprogressive Metastatic Non-Small Cell Lung Cancer or Colorectal Cancer: An Open-Label, Randomized, Controlled Phase 2 Study
Brief Title: 125I Seed Implantation Plus Systemic Therapy for Oligoprogressive NSCLC or Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Li Min (Other)
Responsible Party: Sponsor-Investigator, Li Min, Vice Director, Jinan Military General Hospital
Organization: Jinan Military General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960HP20251214
Record Dates: First submitted 2025-12-16; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Oligometastatic Disease
Keywords: lodine-125 Seed Brachytherapy; Oligoprogression; Non-Small Cell Lung Cancer; Colorectal Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-assignment, open-label interventional study comparing standard-of-care systemic therapy alone with image-guided 125I seed implantation plus standard-of-care systemic therapy in patients with oligoprogressive metastatic non-small cell lung cancer or colorectal cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): Participants receive standard-of-care systemic anticancer therapy per treating physician discretion, which may include chemotherapy, immunotherapy, targeted therapy, and/or maintenance therapy according to current clinical guidelines and individual molecular profiles.
  Interventions: Other: Standard-of-Care Systemic Therapy
- 125I Seed Implantation plus Standard of Care (Experimental): Participants undergo image-guided 125I seed implantation to all extracranial oligoprogressive lesions, followed by continuation of standard-of-care systemic anticancer therapy as determined by the treating physician.
  Interventions: Other: Standard-of-Care Systemic Therapy; Procedure: 125I Seed Implantation

INTERVENTIONS:
Other: Standard-of-Care Systemic Therapy — Standard systemic anticancer therapy administered according to current clinical guidelines and treating physician discretion, which may include chemotherapy, immunotherapy, targeted therapy, and/or maintenance therapy.
Procedure: 125I Seed Implantation — Image-guided implantation of iodine-125 (125I) radioactive seeds to all extracranial oligoprogressive lesions for local tumor control, performed under CT or PET/CT guidance according to institutional standards.
  Arms: 125I Seed Implantation plus Standard of Care

SUMMARY:
Most patients with metastatic cancer eventually develop resistance to systemic therapy. A subset of patients experience oligoprogression, characterized by progression at a limited number of lesions while other disease sites remain controlled by ongoing systemic therapy. This randomized phase 2 trial evaluates whether image-guided 125I seed implantation targeting all oligoprogressive extracranial lesions, combined with standard-of-care systemic therapy, improves progression-free survival compared with standard-of-care systemic therapy alone in patients with metastatic NSCLC or CRC.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized phase 2 controlled trial enrolling adults with histologically confirmed metastatic NSCLC or colorectal cancer who developed extracranial oligoprogression (≤5 progressive lesions) on PET/CT or CT while receiving at least first-line systemic therapy (including maintenance). Eligible patients will be randomized 1:1 to (1) standard-of-care systemic therapy per treating physician discretion, or (2) image-guided 125I seed implantation to all oligoprogressive lesions plus standard-of-care systemic therapy.

Oligoprogression will be determined by predefined imaging response criteria (RECIST and/or PERCIST, depending on baseline imaging modality), with confirmation by designated study radiologists. Follow-up imaging will be performed at 8 weeks (±2 weeks) after randomization and every 12 weeks (±2 weeks) thereafter to assess disease status. The primary endpoint is progression-free survival measured up to 12 months. Secondary endpoints include overall survival, time to initiation of a new systemic therapy, local control of implanted lesions, safety, and quality of life. Optional exploratory objectives may include circulating tumor DNA dynamics and metabolic PET parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically or cytologically confirmed metastatic non-small cell lung cancer (NSCLC) or colorectal cancer (CRC).
* Presence of metastatic disease with extracranial oligoprogression, defined as progression in up to five (≤5) individual lesions on CT or PET/CT imaging, while other known disease sites remain stable or controlled.
* Received at least one prior line of standard systemic anticancer therapy, including maintenance therapy, for metastatic disease.
* All oligoprogressive lesions are technically feasible and considered safe for image-guided 125I seed implantation, as determined by the treating interventional team.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2. Adequate organ function to undergo interventional procedures and systemic therapy, per institutional standards.
* Ability to understand and willingness to sign written informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Leptomeningeal disease or diffuse central nervous system involvement. Uncontrolled infection or serious medical comorbidities that, in the investigator's judgment, would preclude safe participation or interventional procedures.
* Prior radiotherapy or brachytherapy requiring re-irradiation to the same tumor location planned for 125I seed implantation.
* Known bleeding diathesis or uncorrectable coagulation disorders contraindicating interventional procedures.
* Any other condition that, in the investigator's judgment, would make the patient unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From randomization up to 12 months
  Progression-free survival is defined as the time from randomization to systemic disease progression or death from any cause, whichever occurs first. Disease progression will be assessed using RECIST version 1.1 and/or PERCIST criteria based on the baseline imaging modality.

SECONDARY OUTCOMES:
Overall Survival (OS) | From randomization up to 24 months
  Overall survival is defined as the time from randomization to death from any cause.
Time to Initiation of a New Systemic Therapy (TTNT) | From randomization up to 12 months
  Time to initiation of a new systemic therapy is defined as the time from randomization to the start of a new line or regimen of systemic anticancer therapy due to disease progression or clinical decision.
Local Control of Treated Lesions | From intervention to 12 months after randomization
  Local control is defined as the absence of in-field progression of oligoprogressive lesions treated with 125I seed implantation, assessed on follow-up imaging.
Safety and Treatment-Related Adverse Events | From intervention through 12 months
  Safety is assessed by the incidence and severity of adverse events, including procedure-related toxicities, graded according to the Common Terminology Criteria for Adverse Events (CTCAE).

OTHER OUTCOMES:
Metabolic Response on PET Imaging | Baseline and first scheduled imaging assessment (approximately 8 weeks after randomization)
  Metabolic response on PET imaging is defined as the change from baseline in maximum standardized uptake value (SUVmax) of the target lesion, as measured on PET imaging at baseline and follow-up.
Patterns of Disease Progression | From the date of randomization until the date of first documented disease progression, assessed up to 24 months.
  Patterns of disease progression will be descriptively analyzed, including the development of new metastatic lesions versus progression of pre-existing lesions, based on radiographic and/or clinical assessment at the time of disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Min Li, M.D., Study Director — The 960th Hospital of People's Liberation Army (PLA)
Locations (1):
- The 960th Hospital of People's Liberation Army (PLA), Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be made available to qualified researchers upon reasonable request after completion of the study and publication of the primary results. Data to be shared may include demographic information, treatment assignment, key efficacy outcomes, adverse events, and imaging-derived parameters. A data-sharing agreement will be required to ensure appropriate use of the dataset.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following publication, or until the main study database is closed, whichever occurs first.
Access Criteria: Qualified researchers affiliated with academic institutions or recognized research organizations may request access to de-identified individual participant data (IPD), including imaging-derived parameters, dosimetric results, and clinical outcome data.
  Requests must include a brief research proposal describing the scientific rationale, objectives, and planned analyses. Approval will be granted by the study's principal investigator and institutional ethics committee. Data will be shared through secure institutional data transfer systems after execution of a formal data sharing agreement that ensures patient confidentiality and compliance with applicable privacy regulations.